CLINICAL TRIAL: NCT05328778
Title: Pharmacokinetics of Sugammadex in Reversal of Vecuronium-induced Neuromuscular Blockade in Patients During Laparoscopic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, Clinical Professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Laparoscopic Surgery
Record Dates: First submitted 2022-03-04; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pharmacokinetics
Keywords: Sugammadex; Laparoscopic Surgery
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Normal Weight group (Experimental): n=16, 18.5kg/m² ≤ BMI ≤ 24.9kg/m²
  Interventions: Drug: Sugammadex
- Obese group (Experimental): n=16, 25≤BMI≤39.9kg/m²
  Interventions: Drug: Sugammadex
- Morbidly Obese group (Experimental): n=16, BMI≥40kg/m²
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Each patient received a single dose administration of sugammadex 2mg/kg according to the ideal body weight (IBW) at reappearance of the second twitch of the train-of-four (TOF).
  Other Names: Bridion; Org 25969

SUMMARY:
The purpose of this study is to illustrate pharmacokinetics of sugammadex in reversal of vecuronium-induced neuromuscular blockade in patients during laparoscopic surgery

DETAILED DESCRIPTION:
48 patients undergoing laparoscopic surgery were divided into 3 groups according to body mass index (BMI), including normal weight group(A group,n=16,18.5kg/m² ≤ BMI ≤ 24.9kg/m²),obese group (B group, n=16, 25≤BMI≤39.9kg/m²) and morbidly obese group (C group, n=16, BMI≥40kg/m²).

Vecuronium was continuous infusing to maintain moderate neuromuscular blockade during the laparoscopic surgery and stopped infusing after the laparoscopic procedure. A single dose administration of sugammadex (Sug) 2.0mg/kg according to ideal body weight (IBW) was given at the reappearance of the second twitch of the train-of-four (TOF) response.

On one hand, venous blood samples were obtained before administration of Sug and at 2, 3, 5, 10, 15, 20, 30, 60 minutes and 2, 4, 6, 8 hours after administration of Sug to determine plasma concentration of Sug using HPLC-MS. On the other hand, time from start of administration of Sug to recovery of TOF ratio to 0.9 and other clinical indicators were also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. ASA: Ⅰ~Ⅲ
2. BMI≥25kg/m²
3. Patients receiving bariatric surgery.

Exclusion Criteria:

1. Pregnant or lactating women
2. Neuromuscular diseases
3. Malignant hyperthermia or allergic history during general anesthesia
4. Drugs that react with rocuronium and vecuronium were taken

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Sugammadex | 0, 2, 3, 5, 10, 15, 20, 30, 60 minutes and 2, 4, 6, 8 hours
  venous blood samples were obtained
TOF ratio of Recovery Time | TOF ratio at 30, 60, 90, 120, 150 seconds after administration
  time from start of administration of Sug to recovery of TOF ratio to 0.9 and other indicators

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China